CLINICAL TRIAL: NCT04476420
Title: Comparison of Nigella Sativa Oil With Conventional Management on Clinical Outcomes in Oral Submucous Fibrosis
Brief Title: Comparative Effect of Nigella Sativa and Conventional Management for OSMF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Hira Batool, Doctor, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2130520HBOM
Record Dates: First submitted 2020-07-02; First posted 2020-07-20 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Oral Submucous Fibrosis
Keywords: OSMF
MeSH Terms: conditions — Oral Submucous Fibrosis | interventions — Nigella sativa oil; Betamethasone Valerate; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid group (Active Comparator): Participants in group 1 will be given corticosteroid lotion (Betamethasone valerate 0.1%) and will be advised to apply it topically (0.5 ml) on the buccal mucosa thrice a day along with physiotherapy using ice cream sticks three times a day for the duration of 10 minutes (3-5minutes on each side).
  Interventions: Drug: Betamethasone Valerate
- Nigella Sativa oil group (Experimental): Group 2 will be given commercially available, cold pressed N.sativa (Black seed) oil and will be advised to apply it topically over the buccal mucosa (1 ml) thrice a day along with physiotherapy using ice cream sticks three times a day for the duration of 10 minutes (3-5minutes on each side).
  Interventions: Dietary Supplement: Nigella sativa oil

INTERVENTIONS:
Dietary Supplement: Nigella sativa oil — Using N.sativa oil as an alternative to conventional management will help us to find a treatment option which is non-invasive, cost effective, inexpensive, easy available and belongs to a natural source with almost no side effects.
  Arms: Nigella Sativa oil group
Drug: Betamethasone Valerate — it is a conventionally used drug for treating OSMF
  Other Names: Corticosteroid
  Arms: Steroid group

SUMMARY:
Oral submucous fibrosis (OSMF) is a potentially malignant condition mainly characterized by inflammation and fibrosis of the submucosal tissues leading to marked rigidity and reduced opening of the jaws. OSMF has a multifactorial etiology but areca nut consumption is considered to be the most consistent factor in its pathogenesis. There is no definitive treatment available for treating OSMF. Conventional management involves physiotherapy exercises and treating the disease with certain medications such as steroids and homeopathic medications.

DETAILED DESCRIPTION:
OSMF is a chronic insidious disorder of the oral cavity which has a great potential to turn malignant. The clinical manifestations of OSMF comprise of white, marble-like appearance of the oral mucosa with loss of flexibility and formation of palpable fibrous bands extending from the anterior to the posterior region of the oral cavity.Other features include burning sensation on taking spicy food, loss of papillae of the tongue, loss of natural pigmentation of the lips and restricted mouth opening.

There is no definitive treatment available for OSMF due to its complex etiology. The most essential component in the management of OSMF is the discontinuation of the habit of areca nut chewing by the patient followed by conservative or surgical treatment. Currently, steroids are the most commonly used drug group in managing OSMF because of their ability to reduce the inflammatory process and increasing the apoptosis of inflammatory cells thereby decreasing fibrosis. However, they are not very useful in reversing the pathology and restoring mucosal elasticity and can cause mucosal thinning with long term use ultimately resulting in worsening of the symptoms of the disease.

Many in- vitro and in- vivo studies have been conducted to establish the anti neoplastic, anti inflammatory, immunomodulatory, antihypertensive, antimicrobial, anti-parasitic, antioxidant and hypoglycemic properties of N.sativa oil. Among all the constituents of Nigella sativa, Thymoquinone (Tq) is the most pharmacologically active constituent responsible for most of its properties. Nigella sativa has been used widely in different food preparations in the form of a flavoring agent or a spice. It is also recognized as 'safe' in the inventory of United States Food and Drug administration.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the age of 18 years and above
* Patients clinically diagnosed with Oral submucous fibrosis
* Patients who have not received any treatment for Oral submucous fibrosis in the last three months.
* Patients who are willing to quit the habit of eating pan, gutka and areca nut
* Patients who are willing to attend the follow up visits

Exclusion Criteria:

* Patients who are less than 18 years of age
* Patients who are already using pain medications, corticosteroids or immunosuppressive drugs in any other form
* Patients with a history of malignancy
* Patients presenting with oral lesions other than Oral submucous fibrosis (OSMF)
* Patients who are allergic to the drug material used in the clinical trial
* Patients who will not give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-02-11 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Pain assessed using visual analogue scale (VAS) | 6 months
  Pain will be measured using VAS. This scale usually present as a 100-mm horizontal line on which the pain intensity experienced by the patient will be represented by a point between the extremes of "no pain at all" and "worst pain imaginable.
Inter-incisal mouth opening (IMO) assessed using vernier caliper | 6 months
  Interincisal mouth opening will be calculated by measuring the distance between the mesioincisal angles of the maxillary central incisor and the mandibular central incisor with the help of a vernier calliper.

SECONDARY OUTCOMES:
Cheek Flexibility assessed following the method of Mathur and Jha (1993) | 6 months
  A line will be drawn from the tragus of the ear to the angle of the mouth and then two reference points will be marked on both the cheeks at 1/3rd the distance from the angle of the mouth on the line drawn previously. After marking these reference points, the patient will be asked to blow his cheek and the distance will be measured between the two points. Then the patient will be instructed to relax his cheeks and the distance will be measured again. The difference between the two values will give the value for cheek flexibility.
Tongue protrusion | 6 months
  Tongue protrusion will be recorded by measuring the distance between the tip of the tongue and the mesioincisal angle of the upper central incisor using steel ruler.

CONTACTS AND LOCATIONS:
Overall Officials: Hira Batool, Mphil, Principal Investigator — Ziauddin University
Locations (1):
- Ziauddin University, Clifton, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No